CLINICAL TRIAL: NCT04344522
Title: Descemet Membrane Endothelial Keratoplasty Combined With Intraocular Lens Exchange: Sequential Versus Combined Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Kolaib, Ophthalmology resident, Alexandria University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DMEK ACIOL
Record Dates: First submitted 2020-04-03; First posted 2020-04-14 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Pseudophakic Bullous Keratopathy; Anterior Chamber Intraocular Lens
Keywords: Descemet membrane endothelial keratoplasty DMEK; Anterior chamber intraocular lens AC IOL; pseudophakic bullous keratopathy PBK

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- sequential 2 stage procedure (Experimental): In this arm , the procedure will be performed in two stages ; the first stage will include performing IOL exchange together with iridoplasty ( if required) and inferior peripheral iridectomy (PI) and the second stage is performing DMEK one month later
  Interventions: Procedure: Descemet membrane endothelial keratoplasty DMEK; Procedure: IOL exchange; Procedure: iridoplasty; Procedure: Inferior peripheral iridectomy
- combined single stage procedure (Experimental): In this arm, both IOL exchange and DMEK will be performed in the same setting
  Interventions: Procedure: Descemet membrane endothelial keratoplasty DMEK; Procedure: IOL exchange; Procedure: iridoplasty; Procedure: Inferior peripheral iridectomy

INTERVENTIONS:
Procedure: Descemet membrane endothelial keratoplasty DMEK — DMEK : it involves separating the Descemet membrane from a corneal donor graft , doing a descematorhexis in the recepient cornea , loading and injection of the graft into the anterior chamber , unfolding and fixing the graft to the recepient cornea by intracameral air bubble.
Procedure: IOL exchange — IOL exchange : it involves performing a corneoscleral tunnel , freeing the AC IOL from any adhesions and explanting it through the tunnel , then implanting a posterior chamber PMMA lens or iris claw lens if there is no adequate capsular support.
Procedure: iridoplasty — iridoplasty : repairing any iris defect by using 10/0 prolene.
Procedure: Inferior peripheral iridectomy — Inferior peripheral iridectomy : performed by vannus scissor to avoid postoperative pupillary block due to the intracameral air .

SUMMARY:
Surgical treatment of corneal endothelial decompensation in the presence of an anterior chamber intraocular lens (AC IOL) is technically challenging. The ultimate management is to perform Descemet membrane endothelial keratoplasty (DMEK). However , unfolding the DMEK graft in the presence of an AC IOL can be difficult and injurious to the graft so the investigators recommend exchanging the AC IOL with a posterior chamber IOL first. In this study , the investigators aim to compare the outcome and complications of performing DMEK and IOL exchange as combined one stage surgery versus .sequential 2 stage procedure

DETAILED DESCRIPTION:
Pseudophakic Bullous keratopathy is the second leading indication for endothelial keratoplasty. One of the main controversies in the management of PBK in the presence of an AC IOl is whether to retain the IOL or perform an IOL exchange with a PC IOL. The investigators believe that retention of an AC IOL can be hazardous to the DMEK graft due to reduced depth of the anterior chamber and traumatic touch between the graft and the IOL during graft unfolding and even postoperatively. On the other hand , performing an IOL exchange is relatively time consuming and requires excess manipulation of the iris tissue with the risk of intraoperative hyphema and postoperative inflammation which can affect the endothelial graft survival and cell count.

Aim of the study : to compare the outcome and complications between performing intraocular lens (IOL) exchange and Descemet membrane endothelial keratoplasty (DMEK) as single stage versus two stage procedure in the management of pseudophakic bullous keratopathy associated with anterior chamber IOL.

Methods :

The study will be a prospective randomized controlled trial. Eligible subjects with pseudophakic bullous keratopathy and AC IOL will be assigned into two groups each comprising 10 eyes. One group will undergo AC IOL exchange with posterior chamber (PC) IOL ( Poly methyl methacrylate (PMMA) lens or iris claw lens if there is no adequate capsular support) combined with DMEK in the same setting. The other group will undergo 2 stage procedure ; first one is IOL exchange , iridoplasty (if required) and inferior peripheral iridectomy and the second stage is DMEK one month later.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having pseudophakic bullous keratopathy associated with an anterior chamber intraocular lens.
2. Age above 18 years old.

Exclusion Criteria:

1. Patients with corneal stromal scarring .
2. Patients who had prior glaucoma drainage devices implantation. 3 Patient with non-repairable loss in the iris tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
postoperative endothelial cell loss in percentage | 3 months
  The postoperative endothelial cell count will be determined in cell/mm2 using the Konan Cellchek specular microscope (Konan Medical , Irvine, California , USA) at 3 months and compared to the preoperative endothelial cell count of the donor graft to calculate the percentage of endothelial cell loss
Best spectacle corrected visual acuity | 3 months
  best spectacle corrected visual acuity using the decimal system
postoperative hyphema and and intraocular pressure spikes | 1month postoperatively
  Any postoperative hyphema and anterior chamber inflammatory reactions will determined by slit lamp examination:
  Hyphema if found will be graded into :
  1. Microscopic hyphema : circulating red blood cells in the AC
  2. Grade I : less than one third the AC
  3. Grade II: one third to one half the AC
  4. Grade III: more than one half the AC but not total
  5. Grade IV : total hyphema. and intraocular pressure spikes will detected using the Goldmann applanation tonometer to measure the intraocular pressure in mmHg
Postoperative AC inflammatory reactions | 1 month postoperatively
  postoperative AC inflammatory reactions including cell and flare will be determined by slit lamp examination under high magnification:
  AC cells will be graded according to the Standardization of Uveitis Nomenclature (SUN) group grading system as following :
  Grade 0 : 5 or less cells in 1*1mm slit beam Grade 1 : 6- 15 cells in 1*1mm slit beam Grade II : 16-25 cells in 1*1mm slit beam Grade III : 26-50 cells in 1*1mm slit beam grade IV : more than 50 cells in 1*1mm slit beam .
  AC flare will be graded according to the SUN grading system :
  Grade 0 : none Grade I : faint Grade II : moderate ( iris and lens details still seen ) Grade III : Marked ( iris and lens details hazy) Grade IV : intense ( fixed and plastic aqueous ).
Postoperative intraocular pressure spikes | 1 month postoperatively
  postoperative intracular pressure will be measured by Goldmann Applanation Tonometer in mmHg

SECONDARY OUTCOMES:
Keratometric values | 3 months
  Keratometric values will be determined in Diopters using Autorefractometer/Keratometer , the difference between the steep and flat keratometric values will determine the corneal astigamtism in diopters
central corneal thickness | 3 months postoperatively
  central corneal thickness will be determined in micrometer using the Konan Cellchek specular microscope (Konan Medical , Irvine, California , USA)
graft detachment | 1 week postoperatively
  The occurrence of postoperative graft detachment will be determined by slit lamp examination . The incidence of graft detachment will be determined in each group .
Spherical equivalent | 3 months postoperatively
  spherical equivalent will be determined using the autorefractometer in diopters

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Kolaib, MBBCh, Principal Investigator — Alexandria Faculty of Medicine; Mohamed B Goweida, MD, Study Chair — Alexandria Faculty of Medicine
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melles GR, Ong TS, Ververs B, van der Wees J. Preliminary clinical results of Descemet membrane endothelial keratoplasty. Am J Ophthalmol. 2008 Feb;145(2):222-227. doi: 10.1016/j.ajo.2007.09.021. Epub 2007 Dec 3. PMID 18061137
- [Background] Ham L, Dapena I, van Luijk C, van der Wees J, Melles GR. Descemet membrane endothelial keratoplasty (DMEK) for Fuchs endothelial dystrophy: review of the first 50 consecutive cases. Eye (Lond). 2009 Oct;23(10):1990-8. doi: 10.1038/eye.2008.393. Epub 2009 Jan 30. PMID 19182768
- [Background] Dapena I, Ham L, Melles GR. Endothelial keratoplasty: DSEK/DSAEK or DMEK--the thinner the better? Curr Opin Ophthalmol. 2009 Jul;20(4):299-307. doi: 10.1097/ICU.0b013e32832b8d18. PMID 19417653
- [Background] Woo JH, Ang M, Htoon HM, Tan D. Descemet Membrane Endothelial Keratoplasty Versus Descemet Stripping Automated Endothelial Keratoplasty and Penetrating Keratoplasty. Am J Ophthalmol. 2019 Nov;207:288-303. doi: 10.1016/j.ajo.2019.06.012. Epub 2019 Jun 19. PMID 31228467
- [Background] Pricopie S, Istrate S, Voinea L, Leasu C, Paun V, Radu C. Pseudophakic bullous keratopathy. Rom J Ophthalmol. 2017 Apr-Jun;61(2):90-94. doi: 10.22336/rjo.2017.17. PMID 29450379
- [Background] Ravalico G, Botteri E, Baccara F. Long-term endothelial changes after implantation of anterior chamber intraocular lenses in cataract surgery. J Cataract Refract Surg. 2003 Oct;29(10):1918-23. doi: 10.1016/s0886-3350(02)02052-7. PMID 14604711
- [Background] Liarakos VS, Ham L, Dapena I, Tong CM, Quilendrino R, Yeh RY, Melles GR. Endothelial keratoplasty for bullous keratopathy in eyes with an anterior chamber intraocular lens. J Cataract Refract Surg. 2013 Dec;39(12):1835-45. doi: 10.1016/j.jcrs.2013.05.045. PMID 24286840
- [Background] Gupta PK, Bordelon A, Vroman DT, Afshari NA, Kim T. Early outcomes of descemet stripping automated endothelial keratoplasty in pseudophakic eyes with anterior chamber intraocular lenses. Am J Ophthalmol. 2011 Jan;151(1):24-28.e1. doi: 10.1016/j.ajo.2010.07.003. Epub 2010 Oct 20. PMID 20970110